CLINICAL TRIAL: NCT04969627
Title: Effects of GLP-1 Analogue Combined With Metformin and Metformin on Gonadal and Metabolic Profiles in Chinese Overweight/Obese PCOS Patients With Hyperandrogenemia.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bing He (Other)
Responsible Party: Sponsor-Investigator, Bing He, Professor, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020PS624K
Record Dates: First submitted 2021-03-22; First posted 2021-07-21 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Metformin (BMI<24) (Active Comparator): Subjects: PCOS patients whoseBMI<24 Drug: Glucophage Generic name: Metformin Dosage form: 500mg Dosage: 1500-2000mg/day Frequency: 500mg three times a day/1000mg twice a day Duration: 3 months
  Interventions: Drug: Metformin
- Metformin (BMI≥24) (Experimental): Subjects: PCOS patients whoseBMI≥24 Drug: Glucophage Generic name: Metformin Dosage form: 500mg Dosage: 1500-2000mg/day Frequency: 500mg three times a day/1000mg twice a day Duration: 3 months
  Interventions: Drug: Metformin
- Combination (BMI<24) (Experimental): Subjects: PCOS patients whoseBMI<24 Drug: Byetta and Glucophage Generic name: Exenatide Dosage form: Exenatide 5ug and 10ug; Metformin 500mg Dosage: Exenatide10-20ug/day; Metformin 1500-2000mg/day Frequency: Exenatide twice a day; Metformin 500mg three times a day/1000mg twice a day Duration: 3 months
  Interventions: Drug: Metformin; Drug: Exenatide
- Combination (BMI≥24) (Experimental): Subjects: PCOS patients whoseBMI≥24 Drug: Byetta and Glucophage Generic name: Exenatide Dosage form: Exenatide 5ug and 10ug; Metformin 500mg Dosage: Exenatide10-20ug/day; Metformin 1500-2000mg/day Frequency: Exenatide twice a day; Metformin 500mg three times a day/1000mg twice a day Duration: 3 months
  Interventions: Drug: Metformin; Drug: Exenatide

INTERVENTIONS:
Drug: Metformin — Use Metformin for 3 months to treat PCOS
Drug: Exenatide — Use Exenatide for 3 months to treat PCOS
  Arms: Combination (BMI<24); Combination (BMI≥24)

SUMMARY:
To study the effects of GLP-1 analogues combined with metformin and metformin on gonadal and metabolic profiles in PCOS patients with BMI ≥ 24 in China. 60 cases of overweight PCOS patients were collected from Shengjing hospital. The intervention period was 3 months after intervention with met or met + GLP-1. To evaluate the improvement of met or met + GLP-1 in the treatment of hyperandremia, glucose metabolism, BMI, waist circumference, menstruation, hairiness and acne in PCOS patients with different BMI.

ELIGIBILITY:
Inclusion Criteria:

1. Females 18 years to 40 years of age Diagnosed as PCOS by the 2003 Rotterdam criteria
2. Overweight/obesity (BMI≥24 kg/m2)
3. No pregnant plan in recent 6 months
4. Written consent for participation in the study

Exclusion Criteria:

1. type 1 or type 2 diabetes mellitus
2. Subjects have other endocrine diseases, such as adrenal hyperplasias or tumor, androgen-secreting tumors, Cushing's syndrome, thyroid diseases, and hyperprolactinemia
3. Diagnosed with or have a family history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia syndrome type 2 (MEN 2)
4. Serious systemic disease or malignant tumor
5. History of pancreatitis (chronic, acute or recurrent)
6. Body weight change ≥10% at 3 months before treatment
7. Used oral contraceptives or sex hormone drugs in the past 1 month
8. Used oral glucocorticoids in the past 1 month
9. Substance (alcohol or drug) abuse or dependence within 3 months
10. Heavy smokers (smokers who smoke 20 or more cigarettes a day) or heavy drinkers (>10g/d)
11. Subjects have a severe systemic disease, such as cardiovascular system, Renal impairment (eGFR<60ml/min/1.73m2)
12. Increase of transaminases up to < 2.5 times of upper limit of normal value
13. Have a history of thromboembolic disease or thrombotic tendency
14. Subjects in pregnant or lactating or within 1 year after delivery
15. Subjects have an allergic history to the drugs used in the study
16. Subjects have participated in other clinical researches of medicine within 1 month prior to randomization
17. Use of metformin, glucagon-like peptide -1 receptor agonists, or weight loss medications (prescription or OTC) within 30 days before screening

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 60 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Change in body weight | 12 weeks
  Change in body weight

SECONDARY OUTCOMES:
Change in body mass index (BMI) | 12 weeks
  Change in body mass index (BMI)
Change in waist circumference(WC) | 12 weeks
  Change in waist circumference(WC)
Change in Ferriman-Gallwey score | 12 weeks
  Change in Ferriman-Gallwey score，the range of Ferriman-Gallwey score is 0-9, higher scores mean a worse outcome.
Change in Acne severity score | 12 weeks
  Change in Acne severity score,the range of acne severity score is 0-9, higher scores mean a worse outcome.
Changes in frequency of menstrual cycle | 12 weeks
  Changes in frequency of menstrual cycle
Changes in Blood Glucose and Insulin During the oral glucose tolerance test (OGTT) | 12 weeks
  glucose obtained at 0,30,60 and 120 minutes during the OGTT.
Changes in Luteinizing Hormone (LH) | 12 weeks
  Changes in Luteinizing Hormone (LH)
Changes in follicle stimulating hormone (FSH) | 12 weeks
  Changes in follicle stimulating hormone (FSH)
Changes in LH/FSH | 12 weeks
  Changes in LH/FSH
Changes in prolactin (PRL) | 12 weeks
  Changes in prolactin (PRL)
Changes in progesterone (Prog) | 12 weeks
  Changes in progesterone (Prog)
Changes in total testosterone (TT) | 12 weeks
  Changes in total testosterone (TT)
Changes in free testosterone (FT) | 12 weeks
  Changes in free testosterone (FT)
Changes in free androgen index (FAI) | 12 weeks
  Changes in free androgen index (FAI)
Changes in sex hormone binding globulin (SHBG) | 12 weeks
  Changes in sex hormone binding globulin (SHBG)
Changes in dehydroepiandrosterone sulfate (DHEAS) | 12 weeks
  Changes in dehydroepiandrosterone sulfate (DHEAS)
Changes in anti-müllerian hormone (AMH) | 12 weeks
  Changes in anti-müllerian hormone (AMH)

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China